CLINICAL TRIAL: NCT05169541
Title: Is Plasma Level of Mannose Binding Lectin Associated With Reproductive Failure?
Brief Title: Association Between Plasma Level of Mannose Binding Lectin and Human Reproduction
Status: Recruiting | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Caroline Nørgaard-Pedersen, Principal investigator, Aalborg University Hospital
Other Study IDs: MBL_reproduction_2022
Record Dates: First submitted 2021-12-19; First posted 2021-12-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Mannose-Binding Lectin Deficiency; Recurrent Pregnancy Loss; Recurrent Implantation Failure; Infertility; Habitual Abortion; Recurrent Miscarriage; Recurrent Spontaneous Abortion
MeSH Terms: conditions — Mannose-Binding Protein Deficiency; Infertility; Abortion, Habitual; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Recurrent pregnancy loss after spontaneous conception: Minimum three consecutive losses from pregnancies achieved after spontaneous conception
- Recurrent pregnancy loss after assisted reproductive treatment: Minimum three consecutive losses from pregnancies achieved after assisted reproductive treatment (ART), which includes in vitro fertilization (IVF), intracytoplasmic sperm injection (ICSI), and frozen embryo transfer (FER).
- Recurrent implantation failure: Minimum three consecutive embryo transfers (ET) of good quality embryos with no hCG production. The patient must not have experienced any clinical pregnancies (i.e. evidence of pregnancy on an US or by histopathological examination) after IVF or spontaneous conception. Biochemical pregnancies after spontaneous conception, which terminated before evidence of a gestational sac on an ultrasonic scan (US) could be visualized and before the series of RIF occurred, are accepted.

SUMMARY:
A low plasma level of mannose binding lectin (p-MBL) is associated with unexplained recurrent pregnancy loss (RPL), but it is not investigated if it is associated with unexplained reproductive failure in general, including recurrent implantation failure (RIF) after assisted reproductive technology (ART) (including IVF, ICSI and FET), recurrent pregnancy loss (RPL) after spontaneous conception, and RPL after ART.

DETAILED DESCRIPTION:
The prevalence of a low p-MBL level is higher in patients with unexplained RPL than in the background population, while a high level is significantly less frequent in RPL patients (Nørgaard-Pedersen et al., submitted).

Approximately 50% of RPL patients have none of the evidence-based risk factors associated with RPL. Unexplained RPL is more complicated since finding the cause is essential for offering the optimal intervention to improve the patient's chances of a child.

Other conditions characterized by reproductive failure are infertility and recurrent implantation failure (RIF). The underlying mechanisms and the physiologic stage in early pregnancy being complicated and impeding normal pregnancy may probably differ between these pathologic conditions, since theoretically RIF would involve complicated embryo apposition, adhesion and invasion and clinical/visualized pregnancy losses would involve complicated stages later in the implantation process and fetal development. However, these conditions are suggested to have partly overlapping causes since most of the evidence-based risk factor recur; including parental chromosomal abnormalities, and maternal endocrine disorders, acquired thrombophilia, anatomic abnormalities in the uterine cavity, and endometrial and ovarian diseases. In addition, adverse immune responses against the embryo have been suggested as a cause of reproductive failure. If RPL is associated with a low p-MBL level, RIF may be so too.

The investigators aim to explore the p-MBL level in patients suffering from reproductive failure.

If low p-MBL level is associated with all the investigated subgroups of patients suffering from reproductive failure, this would strengthen our theory that MBL is involved in the pathophysiology characterized by reproductive failure in the very early stages of pregnancy and should therefore take part in the exploration of all patients with reproductive failure.

ELIGIBILITY:
Inclusion Criteria:

fulfil one of the following:

* 3 consecutive pregnancy losses after spontaneous conception
* 3 consecutive pregnancy losses after assisted reproductive technology treatment (ART) including IVF, ICSI and FET
* 3 failed embryo transfers characterized by no achieved pregnancy (after 3 cycles with minimum 1 embryo transfer of a good-quality embryo in each cycle.)

Exclusion Criteria:

* Age <18 or >45 years
* AMH <4.0 pmol/l unless donor egg in previous cycles
* Significant uterine malformation
* Known endometrial pathologies including intrauterine endometriosis, adenomyosis, hyperplasia or polyps
* Known chromosomal abnormalities
* Pregnancy >9 weeks of gestation at the time collecting the blood sample

Ages: 18 Years to 41 Years | Sex: Female
Age Groups: Adult
Study Population: Danish female population. The centers cover mainly the western region of Denmark, but patients from all over Denmark can be treated at each center.
  The Aagaard Klinik is a private IVF clinic and therefore their patients pay for their ART treatments. Patients contact the clinic themself when they need medical support because of reproductive failure.
  The RPL center at AaUH (public hospital) is available without costs for the patient. Patients are referred from their practitioner or fertility clinic or gynecologist when they have experienced 3 or more pregnancy losses (including biochemical and clinical pregnancies).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Low p-MBL level | Blood sample collected after admission when the patient is not pregnant or <9 weeks of gestation.
  Low plasma mannose binding lectin level defined as <500 ug/l
Very low p-MBL level | Blood sample collected after admission when the patient is not pregnant or <9 weeks of gestation.
  Very low plasma mannose binding lectin level defined as <100 ug/l
High p-MBL level | Blood sample collected after admission when the patient is not pregnant or <9 weeks of gestation.
  High plasma mannose binding lectin level defined as >3000 ug/l

SECONDARY OUTCOMES:
Odds ratio for a low p-MBL level | Blood sample collected after admission when the patient is not pregnant or <9 weeks of gestation.
  Comparing prevalence in the patient group with danish female background population (n=185)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Nørgaard-Pedersen, M.D., Principal Investigator — Aalborg University Hospital, Denmark
Locations (1):
- Aagaard Klinik, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in RPL after approval by the researchers. Data will be coded with no personal identifiers included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party. Please contact the primary researcher. The researchers maintain the right to reject the request. Data requests can be submitted starting 12 months after article publication.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data requests can be submitted starting 12 months after article publication and up to 36months only on request.
Access Criteria: Only on request.